CLINICAL TRIAL: NCT06199440
Title: Azithromycin Versus Doxycycline on Resistin Level in Periodontitis Patients With Type 2 Diabetes. A Randomized Controlled Clinical Trial
Brief Title: Azithromycin Versus Doxycycline on Restistin Level in Periodontitis Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Jazia Alblowi, Associate Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 121-06-23
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Periodontal Diseases; Type 2 Diabetes
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): Chronic periodontitis patients with diabetes mellitus type II who received scaling and root planning.
  Interventions: Drug: Group I
- Group II (Experimental): Received azithromycin dosage is 250 mg/day for 5 days, after an initial dose of 500 mg one hour before NSPT
  Interventions: Drug: Group II
- Group III (Experimental): Consisted of 5 type 2 Diabetes Mellitus patients with periodontitis who were received doxycycline 20mg twice/day.
  Interventions: Drug: Group III

INTERVENTIONS:
Drug: Group I — First group are chronic periodontitis patients with diabetes mellitus type II who received scaling and root planning.
  Arms: Group I
Drug: Group II — Second group will receive 250 mg of azithromycin per day for a period of 5 days, after an initial dose of 500 mg one hour before NSPT.
  Arms: Group II
Drug: Group III — Third group are Type 2 DM patients who received doxycycline 20mg twice/day.
  Gingival crevicular fluid will be collected at 0, 1, and 3 months to assess Serum Resistin using a human Resistin enzyme-linked immunosorbent assay Kit following the manufacturer's protocol.
  Arms: Group III

SUMMARY:
The aim of this study is to evaluate the adjunctive effects of systemic antibiotics used in nonsurgical periodontal treatment (NSPT), compared with NSPT alone, on the periodontal clinical parameters and resistin level in diabetic patients with periodontitis, in order to identify which, one provides an additional effect to non-surgical periodontal therapy

ELIGIBILITY:
Inclusion Criteria:

Patients were clinically diagnosed as having at least three site with CAL ≥ 5mm; moderate to advanced chronic periodontitis according to the criteria of American Academy of Periodontology.

* Free from any other systemic conditions that affect the periodontium except for Diabetes mellitus type II.
* No periodontal therapy, systemic antibiotics or non-steroidal anti-inflammatory agents during the preceding 6 months.
* Non-smokers.
* Non-pregnant.

Exclusion Criteria:

-

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 3 months
  Improvements in clinical parameters of periodontitis including Gingival Index, Probing Depth and Clinical Attachment Level

SECONDARY OUTCOMES:
Secondary Outcome | 3 months
  Improved resistin level

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No